CLINICAL TRIAL: NCT01986348
Title: A Phase 2 Study Evaluating the Efficacy and Safety of Selinexor (KPT-330) in Patients With Recurrent Gliomas
Brief Title: Study Evaluating the Efficacy and Safety of Selinexor (KPT-330) in Participants With Recurrent Gliomas
Acronym: KING
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to Sponsor decision (all except 1 patient were off-treatment and 2 patients were in survival follow-up)
Sponsor: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCP-330-004
Record Dates: First submitted 2013-10-17; First posted 2013-11-18 (Estimated); Results first posted 2021-08-02 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Glioblastoma; Glioma
Keywords: GBM; Glioblastoma; selinexor; KPT-330; Karyopharm; brain tumor; brain cancer; Glioma; Astrocytoma; Oligodendrogliomas; Oligo-astrocytomas
MeSH Terms: conditions — Glioblastoma; Glioma; Brain Neoplasms; Astrocytoma; Oligodendroglioma | interventions — selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A: Selinexor 60 mg and Surgery (Experimental): Participants who required surgery received up to 3 doses of oral selinexor tablets 60 milligrams (mg) twice weekly (BIW) on Day 1, Day 3 and between 2 and 48 hours prior to surgery, subsequently underwent surgery for resection of their tumor and resumed selinexor tablets 60 mg BIW after recovery, during Week 1 to 4 of each 4-week cycle, until progression of disease (PD) or development of unacceptable toxicities.
  Interventions: Drug: Selinexor
- Arm B: Selinexor 50 mg/m^2 (Experimental): Participants who were not eligible for surgery received selinexor tablets 50 mg per square meter (mg/m^2) BIW during Week 1 to 4 of each 4-week cycle until PD or development of unacceptable toxicities.
  Interventions: Drug: Selinexor
- Arm C: Selinexor 60 mg (Experimental): Participants who were not eligible for surgery received selinexor tablets 60 mg BIW during Week 1 to 4 of each 4-week cycle until PD or development of unacceptable toxicities.
  Interventions: Drug: Selinexor
- Arm D: Selinexor 80 mg (Experimental): Participants who were not eligible for surgery received selinexor tablets 80 mg once weekly (QW) during Week 1 to 4 of each 4-week cycle until PD or development of unacceptable toxicities.
  Interventions: Drug: Selinexor

INTERVENTIONS:
Drug: Selinexor — One cycle is 28 days (4 weeks).
  Other Names: KPT-330

SUMMARY:
This is an open-label, multicenter, Phase 2 study to evaluate the efficacy and safety of oral selinexor in participants with recurrent gliomas.

DETAILED DESCRIPTION:
This is an open-label, multicenter, Phase 2 study to evaluate the efficacy and safety of oral selinexor in participants with recurrent gliomas.

Initially, the study included 2 arms: an exploratory Surgical Arm (Arm A) with sequential enrollment for participants who require surgery and a medical arm (Arm B) for participants who are not eligible for surgery.

Enrollment in Arm B was stopped to explore alternative dosing in Protocol Versions ≥ 4.0 to potentially improve tolerability. Four arms (Arms C, D, E, and F) were added to the Medical Arm in Protocol Version 4.0. Arms E and F were eliminated in protocol version 6.0 and no participants were ever enrolled in these arms.

Participants in the primary population enrolled under Protocol Version ≥ 4.0 will be randomized to Arm C and Arm D (approximately 30 participants per arm) to explore alternative dosing to potentially improve tolerability.

After screening and registration/randomization in the study, participants enrolling in Arm A or randomized to Arm C will receive 60 mg selinexor orally twice weekly. Participants randomized to Arm D will receive 80 mg selinexor orally weekly.

Participants will be treated until progression of disease or the development of unacceptable toxicities. All participants will then undergo the End of Treatment (EOT) visit.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed GBM (including all histologic variants) at first diagnosis with radiographic evidence of recurrent disease after treatment with radiotherapy and temozolomide;
* 18 years of age or older
* Participants enrolling in the medical arm (Arms B, C and D) must be on a stable or decreasing dose of corticosteroids (or none) for at least 5 days prior to the baseline MRI;
* Measurable disease (according to RANO guidelines)
* Surgical arm (Arm A) must be predicted pre-operatively to have sufficiently sized tumor to be resected and provide tissue samples for exploratory assessments.

Exclusion Criteria:

* Markedly decreased visual acuity if attributed to other causes than GBM.
* Known active hepatitis A, B, or C
* Participants with coagulation problems and medically significant bleeding in the month prior to start of treatment (e.g., peptic ulcer, epistaxis, spontaneous bleeding). Prior history of DVT or PE is not exclusionary.
* Participants must not have significantly diseased or obstructed gastrointestinal tract, malabsorption, uncontrolled vomiting or diarrhea, or inability to swallow oral medications.
* Prior treatment with bevacizumab or other direct VEGF/ VEGFR inhibitors. For any question of the definition of a direct VEGF/VEGFR inhibitor, consult Sponsor.
* Arms C and D only: body surface area < 1.2 m².
* < 24 days from prior temozolomide, < 6 weeks from nitrosourea, < 4 weeks from other chemotherapy or investigational agents prior to start of treatment within study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2014-03-03 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-01-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Center for Neuro-Oncology, Boston, Massachusetts
  - Columbia University, Herbert Irving Comprehensive Cancer Center, New York, New York
- The Phase I Unit, Dept. of Oncology, Rigshospitalet, Copenhagen, Denmark
- Netherlands (2):
  - University of Groningen Faculty of Medical Sciences, Medical Oncology, Groningen
  - Erasmus MC-Daniel den Hoed Cancer Center- Neuro-Oncology Unit, Rotterdam

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 6 sites across the United States of America, Denmark and Netherland between 03 March 2014 and 23 January 2020.
Pre-assignment Details: A total of 76 participants were enrolled, randomized and treated in this study.
Period: Overall Study
Arm/Group | Arm A: Selinexor 60 mg and Surgery | Arm B: Selinexor 50 mg/m^2 | Arm C: Selinexor 60 mg | Arm D: Selinexor 80 mg
Started | 8 | 24 | 14 | 30
Completed | 0 | 0 | 0 | 0
Not Completed | 8 | 24 | 14 | 30
Not completed — Death | 8 | 22 | 10 | 21
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Progressive Disease | 0 | 0 | 2 | 0
Not completed — Withdrawal by Participant | 0 | 1 | 2 | 1
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 3
Not completed — Other-unspecified | 0 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety population consisted of all participants who had received any amount of study treatment.
Groups:
- Arm A: Selinexor 60 mg and Surgery: Participants who required surgery received up to 3 doses of oral selinexor tablets 60 mg BIW on Day 1, Day 3 and between 2 and 48 hours prior to surgery, subsequently underwent surgery for resection of their tumor and resumed selinexor tablets 60 mg BIW after recovery, during Week 1 to 4 of each 4-week cycle, until PD or development of unacceptable toxicities.
- Arm B: Selinexor 50 mg/m^2: Participants who were not eligible for surgery received selinexor tablets 50 mg/m^2 BIW during Week 1 to 4 of each 4-week cycle until PD or development of unacceptable toxicities.
- Arm D: Selinexor 80 mg: Participants who were not eligible for surgery received selinexor tablets 80 mg QW during Week 1 to 4 of each 4-week cycle until PD or development of unacceptable toxicities.
- Total: Total of all reporting groups
Arm/Group | Arm A: Selinexor 60 mg and Surgery | Arm B: Selinexor 50 mg/m^2 | Arm C: Selinexor 60 mg | Arm D: Selinexor 80 mg | Total
Number analyzed (Participants) | 8 | 24 | 14 | 30 | 76
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.6 (6.70) | 51.1 (13.04) | 49.5 (12.36) | 54.3 (11.98) | 52.7 (11.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 5 | 11 | 22
  Male | 7 | 19 | 9 | 19 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 3 | 3
  Not Hispanic or Latino | 8 | 20 | 8 | 24 | 60
  Unknown or Not Reported | 0 | 4 | 6 | 3 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 8 | 24 | 8 | 25 | 65
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: 6-Month Progression-Free Survival (PFS) Rate
Description: The analysis of 6mPFS was performed by calculating the estimated survival probability of having PFS ≥ 6 months based on Kaplan-Meier method, where PFS was defined as the time from the start of study treatment until first documented progression based on Response Assessment in Neuro-Oncology (RANO) criteria, or death from any cause. Progressive disease occurs when either of the criteria was present: greater than or equal to (≥) 25 percentage (%) increase in T1 gadolinium enhancing disease, increase in T2/ Fluid-attenuated inversion recovery (FLAIR), detection of new lesions, or decreased clinical status.
Time Frame: From start of study treatment up to disease progression or death, whichever occurred first (assessed up to Month 6)
Population: Modified intent-to-treat (mITT) population consisted of all enrolled participants in Arms B, C and D who had received at least 1 dose of study medication and have at least 1 post-baseline efficacy follow-up assessment, unless the participant discontinued treatment prior to the first post baseline assessment due to death, toxicity, or PD. Data for this outcome measure was not planned to be collected and analyzed for Arm A: Selinexor 60 mg and Surgery.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm B: Selinexor 50 mg/m^2 | Arm C: Selinexor 60 mg | Arm D: Selinexor 80 mg
Number analyzed (Participants) | 24 | 13 | 30
percentage of participants | 9.72 [2.67 to 35.39] | 7.69 [1.17 to 50.57] | 17.24 [7.77 to 38.27]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: The ORR was determined as percentage of participants who had either complete response (CR) or partial response (PR) using the RANO criteria. CR: No T1 gadolinium enhancing disease, stable or decreasing T2/FLAIR, no new lesions, no corticosteroid use and stable, or increasing clinical status. PR: ≥50% decrease in T1 gadolinium enhancing disease, stable or decreasing T2/FLAIR, no new lesions, stable or decreased use of corticosteroids, and stable or increased clinical status.
Time Frame: Up to 71 months
Population: mITT population consisted of all enrolled participants in Arms B, C and D who had received at least 1 dose of study medication and have at least 1 post-baseline efficacy follow-up assessment, unless the participant discontinued treatment prior to the first post baseline assessment due to death, toxicity, or disease progression. Data for this outcome measure was not planned to be collected and analyzed for Arm A: Selinexor 60 mg and Surgery.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm B: Selinexor 50 mg/m^2 | Arm C: Selinexor 60 mg | Arm D: Selinexor 80 mg
Number analyzed (Participants) | 24 | 13 | 30
percentage of participants | 8.3 [1.0 to 27.0] | 7.7 [0.2 to 36.0] | 10.0 [2.1 to 26.5]

3. Secondary Outcome: Overall Survival (OS)
Description: The OS was calculated from the date of start of study treatment to the date of death. Participants who were still alive prior to the data cut-off for final efficacy analysis, or who dropout prior to study end, were censored on the day they were last known to be alive. The OS was estimated using Kaplan-Meier method.
Time Frame: From date of study treatment up to date of death (assessed up to 71 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm B: Selinexor 50 mg/m^2 | Arm C: Selinexor 60 mg | Arm D: Selinexor 80 mg
Number analyzed (Participants) | 24 | 13 | 30
months | 10.51 [4.93 to 16.95] | 8.48 [7.29 to NA] — Data could not be estimated due to higher number (>50%) of censored participants. | 10.15 [7.03 to 15.38]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: The PFS was calculated from the date of start of study treatment to the date of disease progression based on RANO criteria, or date of death should progression not have occurred. Progressive disease occurs when either of the criteria was present: ≥25% increase in T1 gadolinium enhancing disease, increased T2/FLAIR, detection of new lesions, or decreased clinical status.
Time Frame: From start of study treatment up to disease progression (assessed up to 71 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm B: Selinexor 50 mg/m^2 | Arm C: Selinexor 60 mg | Arm D: Selinexor 80 mg
Number analyzed (Participants) | 24 | 13 | 30
months | 1.64 [1.18 to 3.15] | 1.87 [1.84 to 14.88] | 1.87 [1.81 to 3.02]

5. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. A serious adverse event (SAE) was defined as an AE that was fatal; life threatening (places the participant at immediate risk of death); requires in-patient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; was a congenital anomaly/birth defect; and other important medical events. TEAE was defined as any AE with onset or worsening of a pre-existing condition on or after the first administration of study medication through 30 days following last dose or any event considered drug-related by the Investigator through the end of the study. TEAEs included both serious and non-serious TEAEs.
Time Frame: From start of study treatment administration up to 71 months
Population: Safety population consisted of all participants who had received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Selinexor 60 mg and Surgery | Arm B: Selinexor 50 mg/m^2 | Arm C: Selinexor 60 mg | Arm D: Selinexor 80 mg
Number analyzed (Participants) | 8 | 24 | 14 | 30
Participants
  Participants with TEAEs | 8 | 24 | 14 | 30
  Participants with TESAEs | 5 | 7 | 7 | 7

ADVERSE EVENTS:
Time Frame: From start of study treatment administration up to 71 months
Arm/Group | Arm A: Selinexor 60 mg and Surgery | Arm B: Selinexor 50 mg/m^2 | Arm C: Selinexor 60 mg | Arm D: Selinexor 80 mg
All-Cause Mortality (participants affected / at risk) | 8/8 | 22/24 | 10/14 | 21/30
Serious Adverse Events (participants affected / at risk) | 5/8 | 7/24 | 7/14 | 7/30
Other Adverse Events (participants affected / at risk) | 8/8 | 24/24 | 14/14 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Selinexor 60 mg and Surgery (N=8) | Arm B: Selinexor 50 mg/m^2 (N=24) | Arm C: Selinexor 60 mg (N=14) | Arm D: Selinexor 80 mg (N=30)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2
Meningitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Shunt malfunction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 3 | 2
Syncope (Nervous system disorders) | 0 | 0 | 0 | 3
Headache (Nervous system disorders) | 0 | 1 | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Pneumocephalus (Nervous system disorders) | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Embolism (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Selinexor 60 mg and Surgery (N=8) | Arm B: Selinexor 50 mg/m^2 (N=24) | Arm C: Selinexor 60 mg (N=14) | Arm D: Selinexor 80 mg (N=30)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 16 | 6 | 11
Leukopenia (Blood and lymphatic system disorders) | 0 | 7 | 1 | 14
Neutropenia (Blood and lymphatic system disorders) | 1 | 7 | 2 | 10
Anaemia (Blood and lymphatic system disorders) | 2 | 5 | 1 | 6
Lymphopenia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 8
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 2 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 2
Cushingoid (Endocrine disorders) | 0 | 4 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 6 | 1 | 4
Dry eye (Eye disorders) | 1 | 1 | 1 | 1
Eye pain (Eye disorders) | 1 | 0 | 0 | 2
Periorbital oedema (Eye disorders) | 1 | 1 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 3 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 12 | 9 | 21
Vomiting (Gastrointestinal disorders) | 1 | 9 | 5 | 13
Constipation (Gastrointestinal disorders) | 3 | 8 | 7 | 7
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 3 | 6
Dry mouth (Gastrointestinal disorders) | 1 | 3 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 3
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Fatigue (General disorders) | 5 | 19 | 11 | 16
Gait disturbance (General disorders) | 5 | 5 | 3 | 3
Oedema peripheral (General disorders) | 3 | 1 | 2 | 3
Malaise (General disorders) | 1 | 1 | 3 | 3
Face oedema (General disorders) | 0 | 2 | 2 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 1 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2 | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 5
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Incision site pain (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 5 | 6 | 2
Alanine aminotransferase increased (Investigations) | 2 | 1 | 0 | 5
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0 | 3
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 3 | 12 | 10 | 8
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 11 | 3 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 5 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 4 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 3 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 1
Hyperlipasaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1
Hypercreatininaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hyperamylasaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 3 | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 10 | 6 | 4
Headache (Nervous system disorders) | 4 | 5 | 6 | 5
Dizziness (Nervous system disorders) | 3 | 6 | 4 | 2
Memory impairment (Nervous system disorders) | 1 | 2 | 2 | 2
Aphasia (Nervous system disorders) | 1 | 2 | 0 | 2
Balance disorder (Nervous system disorders) | 1 | 1 | 2 | 1
Dysarthria (Nervous system disorders) | 0 | 4 | 0 | 1
Seizure (Nervous system disorders) | 2 | 1 | 0 | 2
Haemorrhage intracranial (Nervous system disorders) | 2 | 0 | 0 | 2
Hemiparesis (Nervous system disorders) | 1 | 2 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 3 | 0 | 0
Tremor (Nervous system disorders) | 0 | 2 | 0 | 2
Coordination abnormal (Nervous system disorders) | 0 | 2 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 2 | 0 | 0
Hemianopia homonymous (Nervous system disorders) | 0 | 0 | 1 | 1
IIIrd nerve disorder (Nervous system disorders) | 1 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 1
Motor dysfunction (Nervous system disorders) | 0 | 2 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 2
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 2
Visual field defect (Nervous system disorders) | 0 | 1 | 1 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebrospinal fluid leakage (Nervous system disorders) | 1 | 0 | 0 | 0
Intracranial pressure increased (Nervous system disorders) | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
Upper motor neurone lesion (Nervous system disorders) | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 4 | 1 | 5
Depression (Psychiatric disorders) | 1 | 1 | 2 | 1
Insomnia (Psychiatric disorders) | 0 | 4 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 1
Abnormal behaviour (Psychiatric disorders) | 0 | 0 | 2 | 0
Mood altered (Psychiatric disorders) | 0 | 1 | 1 | 0
Personality change (Psychiatric disorders) | 0 | 0 | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 1 | 3 | 2 | 3
Pollakiuria (Renal and urinary disorders) | 0 | 2 | 1 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 6
Flushing (Vascular disorders) | 1 | 1 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 3

LIMITATIONS AND CAVEATS:
Study was terminated due to Sponsor decision (all except 1 patient were off-treatment and 2 patients were in survival follow-up).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2015-11-13): https://cdn.clinicaltrials.gov/large-docs/48/NCT01986348/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-05): https://cdn.clinicaltrials.gov/large-docs/48/NCT01986348/SAP_001.pdf